Long Term Immune Memory Responses to Human Papillomavirus (HPV) Vaccination Following 2 Versus 3 Doses of Quadrivalent HPV Vaccine

(Merck08 Study)

Clinical Trial Registration Number: NCT02968420

**Date:** 15 March 2019

# Data Analysis Plan For Demographic/Clinical Characteristics and Serology Data

**Objective:** To compare the serum antibody responses to HPV 6, 11, 16 and 18 at 7 and 30 days post-booster dose of HPV vaccine in females that received either a primary 2 or 3 dose series of Q-HPV vaccine 8-10 years ago.

**Primary testing** is to determine non-inferiority (95% CI, lower bound >0.5) of geometric mean titer (GMT) ratios for anti-HPV 6, 11, 16, 18 for 2-dose girls compared with 3-dose girls and 3-dose women.

Co-primary endpoints are the antibody levels measured by MERCK using competitive Luminex immunoassay (cLIA) at 7 and 30 days post-booster dose of HPV vaccine.

Co-secondary endpoints are the antibody levels measured by MERCK using total IgG Luminex immunoassay (TIgG) at 7 and 30 days post-booster dose of HPV vaccine. Antibody levels measured by cLIA and TIgG at baseline will also be compared in the three groups.

## **Statistical Analysis:**

## Participation and demographic/clinical Characteristics:

Descriptive analysis (i.e. frequency and/or percentage) will be used to summarize study population, including enrollment, withdraw, loss to follow-up, eligibility (Figure 1); and demographic/clinical characteristics including age, baseline health and immunization history (Table 1).

## **Evaluation of anti-HPV antibody levels:**

Merck employed cLIA and TIgG to measure neutralizing and total IgG antibody response to 9-valent HPV vaccine. To assess anti-HPV antibody levels, we will use the results of cLIA and total IgG at baseline (visit 1), and at 7 days (visit 2) and 30 days (visit 3) post-booster dose of HPV vaccine. GMTs of anti-HPV 6, 11, 16, and 18 antibodies will be computed for each group at the three time points. To allow GMT calculation, samples with undetectable anti-HPV will be assigned the half of the lowest detectable value (*cLIA*: *HPV6*, 2 *mMU/ml*; *HPV11*, 3 *mMU/ml*; *HPV16*, 5 *mMU/ml*; *HPV18*, 10 *mMU/ml*. *TIgG*: Merck08-230

HPV6, 2 mMU/ml; HPV11, 2 mMU/ml; HPV16, 4 mMU/ml; HPV18, 3 mMU/ml). 95% confidence intervals (CIs) of GMT will be calculated by back transformation of the 95% CI for the log-transformed GMT (Table 2-3).

# **Non-inferiority testing:**

To test non-inferiority, t-test will be applied to assess GMT ratios in different groups (2-dose girls vs. 3-dose girls; 2-dose girls vs. 3-dose women; 3-dose girls vs. 3-dose women) at 7 and 30 days post-booster dose of HPV vaccine. Non-inferiority will be declared if the lower bound of the 95% confidence interval (95% CI) of GMT ratios is greater than 0.5 (Table 2-3).

#### **Evaluation of seropositivity:**

Seropositivity will be examined for the three groups at baseline, and at 7 and 30 days post-booster dose of HPV vaccine. Positivity thresholds for cLIA are 20 mMU/mL, 16mMU/mL, 20 mMU/mL, and 24 mMU/mL for anti-HPV 6, 11, 16, and 18, respectively; whereas total IgG 15 mMU/mL, 15mMU/mL, 7 mMU/mL, and 10 mMU/mL respectively. A participant is considered to be seropositive if the respective anti-HPV antibody level exceeds or equal to these threshold (Table 4-5). Chi-squared test will be used to compare seropositivity rate in different groups (2-dose girls vs. 3-dose girls; 2-dose girls vs. 3-dose women; 3-dose girls vs. 3-dose women) at baseline, and at 7 and 30 days post-booster dose of HPV vaccine. A margin of 10% of difference in seropositivity rate will be used for non-inferiority testing.

# Assessment of difference in antibody response over time:

Difference in antibody response over time will be assessed based on log-transformed scale of GMT values at different time points (baseline vs. 7 days; baseline vs. 30 days). Paired t-test will be used to test the difference in each group over time. Two-sample t-test will be used to test difference over time between groups (2-dose girls vs. 3-dose girls; 2-dose girls vs. 3-dose women; 3-dose girls vs. 3-dose women). All of the t-test will be two-sided, at a significant level of 0.05 (Table 6-7).

# **Figures and Tables:**

Figure 1. Study participation consort diagram to summarize enrollment, withdraw, loss of follow-up, eligibility...



Table 1. Demographic/clinical characteristics of the study population

| Characteristics | | Group 1 (2-dose girls) | | oup 2<br>e girls) | Group 3 (3-dose women) | |
|---|---|---|---|---|---|---|
| | N | % | N | % | N | % |
| Age at enrollment, mean (SD), year | | | | | | |
| Age at first dose of Q-HPV vaccine, mea | n (SD), year | | | | | |
| Weight, mean (SD), kg | | | | | | |
| BMI, mean (SD) | | | | | | |
| Ethnicity | | | | | | |
| White | | | | | | |
| Chinese | | | | | | |
| Other | | | | | | |
| Health history | | | | | | |
| Immunization history | | | | | | |

**Group 1**: girls who received 2 doses of Q-HPV vaccine at 0, 6 month schedule 8-10 years ago when they were between 9-13 years of age at the time of the first dose

**Group2**: girls who received 3 doses of Q-HPV vaccine at 0, 2, 6 month schedule 8-10 years ago when they were between 9-13 years of age at the time of the first dose

*Group 3*: young women who received 3 doses of Q-HPV vaccine at 0, 2, 6 month schedule 8-10 years ago when they were between 16-26 years of age at the time of the first dose)

Table 2. Summary of anti-HPV GMTs at baseline, and 7 and 30 days post-booster dose (cLIA)

| Antibodies (cLIA) | Group 1 | (2-dose girls) | Group 2 (3 | 3-dose girls) | Group 3 (3-dose women) | | GMT ratio (95% 0 | | CI) |
|---|---|---|---|---|---|---|---|---|---|
| | n | GMT | n | GMT | n | GMT | 2-dose | 2-dose | 3-dose |
| | | (95% CI) | | (95% CI) | | (95% CI) | girl/3-dose | girl/3-dose | girl/3-dose |
| | | | | | | | girl | women | women |
| | | | | Bas | eline | • | • | | |
| HPV 6 | | | | | | | | | |
| HPV 11 | | | | | | | | | |
| HPV 16 | | | | | | | | | |
| HPV 18 | | | | | | | | | |
| | • | • | | At 7 days pos | t-booster dose | | | | |
| HPV 6 | | | | | | | | | |
| HPV 11 | | | | | | | | | |
| HPV 16 | | | | | | | | | |

| HPV 18 |
|------------------------------|
| At 30 days post-booster dose |
| HPV 6 |
| HPV 11 |
| HPV 16 |
| HPV 18 |

Table 3. Summary of anti-HPV GMTs at baseline, and 7 and 30 days post-booster dose (total IgG)

| Antibodies<br>(IGG) | Group 1 | (2-dose girls) | e girls) Group 2 (3-dose girls) Group 3 (3-dose women) | | GN | GMT ratio (95% CI) | | | |
|---|---|---|---|---|---|---|---|---|---|
| | n | GMT | n | GMT | n | GMT | 2-dose | 2-dose | 3-dose |
| | | (95% CI) | | (95% CI) | | (95% CI) | girl/3-dose | girl/3-dose | girl/3-dose |
| | | | | | | | girl | women | women |
| | I. | <u> </u> | | Bas | eline | L | l | L | L |
| HPV 6 | | | | | | | | | |
| HPV 11 | | | | | | | | | |
| HPV 16 | | | | | | | | | |
| HPV 18 | | | | | | | | | |
| | I. | <u> </u> | | At 7 days pos | st-booster dose | L | l | L | L |
| HPV 6 | | | | | | | | | |
| HPV 11 | | | | | | | | | |
| HPV 16 | | | | | | | | | |
| HPV 18 | | | | | | | | | |
| | l | | | At 30 days po | st-booster dose | ) | l | l . | l . |
| HPV 6 | | | | | | | | | |
| HPV 11 | | | | | | | | | |
| HPV 16 | | | | | | | | | |
| HPV 18 | | | | | | | | | |

Table 4. Summary of HPV seropositivity at baseline, and at 7 and 30 days post-booster dose (cLIA)

| Antibodies (cLIA) | ( | Group 1 (2-dose girls) | Group 2 (3-dose girls) | Group 3 (3-dose women) | |
|---|---|---|---|---|---|
| | n | % seropositive (95% CI) | n % seropositive (95% CI) | | % seropositive (95% CI) |
| | Baseline | | | | |
| HPV 6 | | | | | |
| HPV 11 | | | | | |
| HPV 16 | | | | | |

| HPV 18 | | | | | |
|---|---|---|---|---|---|
| | At 7 days post-booster dose | | | | |
| HPV 6 | | | | | |
| HPV 11 | | | | | |
| HPV 16 | | | | | |
| HPV 18 | | | | | |
| | | At 3 | 0 days po | st-booster dose | • |
| HPV 6 | | | | | |
| HPV 11 | | | | | |
| HPV 16 | | | | | |
| HPV 18 | | | | | |

Table 5. Summary of HPV seropositivity at baseline, and 7 and 30 days post-booster dose (total IGG)

| Antibodies<br>(IGG) | | Group 1 (2-dose girls) | ( | Group 2 (3-dose girls) | G | roup 3 (3-dose women) |
|---|---|---|---|---|---|---|
| | n | % seropositive (95% CI) | n | % seropositive (95% CI) | n | % seropositive (95% CI) |
| | | <u> </u> | Bas | eline | | <u> </u> |
| HPV 6 | | | | | | |
| HPV 11 | | | | | | |
| HPV 16 | | | | | | |
| HPV 18 | | | | | | |
| | | At | 7 days pos | st-booster dose | | I |
| HPV 6 | | | | | | |
| HPV 11 | | | | | | |
| HPV 16 | | | | | | |
| HPV 18 | | | | | | |
| | | At 3 | 0 days po | st-booster dose | | |

6

| HPV 6 |
|--------|
| HPV 11 |
| HPV 16 |
| HPV 18 |

Table 6. Difference in anti- HPV GMTs between baseline vs. at 7 and 30 days post-booster dose of HPV vaccine (cLIA)

| Antibodies | Group 1 (2 | 2-dose | Group 2 (3 | 3-dose | Group 3 ( | 3-dose | Group 1 vs | Group 1 vs | Group 1 vs |
|---|---|---|---|---|---|---|---|---|---|
| (cLIA) | girls | ) | girls | ) | wome | en) | 2 | 3 | 3 |
| | Log<br>Difference | P<br>Value | Log<br>Difference | P<br>value | Log<br>Difference | P value | P-value<br>for<br>difference<br>between<br>differences<br>for group<br>1 vs 2 | P-value for<br>difference<br>between<br>differences<br>for group<br>vs 3 | P-value<br>for<br>difference<br>between<br>differences<br>for group<br>1 vs 3 |
| | | | Baseline vs. 7 | days pos | t-booster dose o | of HPV vacc | eine | <u> </u> | <u> </u> |
| HPV 6 | | | | | | | | | |
| HPV 11 | | | | | | | | | |
| HPV 16 | | | | | | | | | |
| HPV 18 | | | | | | | | | |
| | | | Baseline vs. 3 | 0 days po | st-booster dose | of HPV vac | cine | <u> </u> | |
| HPV 6 | | | | | | | | | |
| HPV 11 | | | | | | | | | |
| HPV 16 | | | | | | | | | |
| HPV 18 | | | | | | | | | |

Table 7. Difference in anti- HPV GMTs between baseline vs. at 7 and 30 days post-booster dose of HPV vaccine (total IgG)

| Antibodies | Group 1 (2 | 2-dose | Group 2 (3-dose | | Group 3 (3-dose | | Group 1 vs | Group 1 vs | Group 1 vs |
|---|---|---|---|---|---|---|---|---|---|
| (IGG) | girls | ) | girls) | | women) | | 2 | 3 | 3 |
| | | | | | | | P-value | P-value for | P-value |
| | Log | P | Log | P | Log | D 1 | for | difference | for |
| | Difference | Value | Difference | value | Difference | P value | difference | between | difference |
| | | | | | | | between | differences | between |
| | | | | | | | differences | for group | differences |

| | | | | | | for group | vs 3 | for group |
|---|---|---|---|---|---|---|---|---|
| | | | | | | 1 vs 2 | | 1 vs 3 |
| | | Baseline vs. 7 | days pos | t-booster dose | of HPV vacc | ine | | |
| HPV 6 | | | | | | | 1 | |
| IIF V O | | | | | | | | |
| HPV 11 | | | | | | | | |
| 111 V 11 | | | | | | | | |
| HPV 16 | | | | | | | | |
| HPV 18 | | | | | | | | |
| l. | I | Baseline vs. 30 | 0 days po | st-booster dos | e of HPV vac | cine | I . | |
| HPV 6 | | | | | | | | |
| HPV 11 | | | | | | | | |
| HPV 16 | | | | | | | | |
| *************************************** | | | | | | | | |
| HPV 18 | | | | | | | | |

Tables for uploading results to ClinicalTrials.gov, as required.